CLINICAL TRIAL: NCT03722797
Title: Metabolic Cost and Physical Activity in Sedentary Adults With a Unilateral Transtibial Amputation as Compared to Controls
Brief Title: Physical Activity in Adults With Amputation
Status: Terminated | Type: Observational
Why Stopped: Equipment used for metabolic testing is no longer serviced and/or supported by the company. Alternative equipment is not available to the research team to continue to conduct the study.
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Jaclyn Sions, Assistant Professor, Department of Physical Therapy, University of Delaware
Other Study IDs: 1046346
Record Dates: First submitted 2018-05-01; First posted 2018-10-29 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Amputees
Keywords: energy metabolism; walking; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral Transtibial Amputation: Individuals with a unilateral, transtibial amputation.
  Interventions: Procedure: Metabolic Cost Testing Procedures
- Controls: Healthy adults without a lower-limb amputation who have been matched to participants in the Unilateral Transtibial Amputation group based on age, sex, and body mass index.
  Interventions: Procedure: Metabolic Cost Testing Procedures

INTERVENTIONS:
Procedure: Metabolic Cost Testing Procedures — The Oxycon Mobile™Portable VO2 Measurement system will be used to measure VO2 uptake during 2 walking tests. Test order will be randomized.
  Treadmill Test: Participants will walk on a treadmill at constant speed, based on the participant's self-selected gait speed, for 2.5 minutes in each stage. Walking will occur at 75% of self-selected gait speed in stage 1, 100% in stage 2, and 125% in stage 3.
  Over-ground Test: Participants will walk in an uncarpeted corridor on a course consisting of 2 cones, 20-meters apart. Participants will be instructed to walk at a constant speed for 2.5 minutes in each stage. Instructions will be to walk at their "slow" speed in stage 1, their "usual, comfortable" speed in stage 2, and their "brisk" speed in stage 3.

SUMMARY:
This cross-sectional study explores physical activity and energy expenditure among inactive adults with a unilateral transtibial amputation. Results may assist with physical activity prescription for adults with unilateral lower-limb loss.

DETAILED DESCRIPTION:
Up to 48% of adults following a lower-limb amputation will die within the upcoming year. Lack of physical activity (exercise) contributes to high death rates. It is recommended that younger (and middle-aged) adults without a health condition walk 10,000 steps/day to reduce the risk of chronic health conditions, while recommendations are 7,100 steps per day for older adults and those with chronic health conditions. Adults with a lower-limb amputation walking about 21-43% of the recommended 7,100 steps/day. Step activity monitors, such as the StepWatch (a research-grade accelerometer) and the FitBit (a commercially-available monitor) provide a means of evaluating physical activity, which is important since patients tend to over-estimate their level of physical activity. Activity monitor use, however, may not be possible in every healthcare practice setting, as monitors may cost $100-$600 and someone must remove the data from the monitor, interpret the data, and enter the data into the patient's medical record. Therefore, physical activity questionnaires, where the patient self-reports their physical activity, are ideal in a clinical setting. Unfortunately, to date, there has been little research looking at the accuracy of physical activity questionnaires in patients with lower-limb amputations and how these questionnaires measure up to data obtained from step activity monitors.

In addition to 7,100 steps/day, adults with mobility-limiting, chronic conditions (including individuals with lower-limb amputations) should participate in ≥150 minutes of moderate-intensity physical activity per week, with activity in ≥10 minutes per bout. Moderate-intensity activity has been defined as 3 metabolic equivalents (METs). One MET is equal to the amount of oxygen one consumes at rest, so 3 METs means that one is consuming 3 times the amount of oxygen one would consume at rest. In healthy adults without a medical condition this equates to walking 2.6-2.7 mph or 100 steps/minute, while for adults with an amputation of the leg below-the-knee (i.e. a transtibial amputation), 1.47 mph or 86 steps/minute has been reported to equal 3 METs. Maximal walking speeds for adults with lower-limb amputations, specifically those who have lost their limb due to poor blood circulation may be ≤1.67 mph, so one must question if walking 1.47 mph for an extended time is possible for these patients. Investigators believe that 1.47mph is greater than 3 METs for adults with a lower-limb amputation who have other medical issues, such as diabetes and peripheral vascular disease, and who are deconditioned and not participating in physical activity.

It is important to know what speed (mph) and cadence (steps/minute) equals 3 METs in adults with a lower-limb amputation with other medical conditions who are currently inactive. Investigators believe that these patients represent the vast majority of patients that healthcare providers encounter and must council regarding increasing physical activity levels. Providers need to know what speed and cadence is equal to 3 METs for inactive patients with limb loss with other medical conditions, so that providers can appropriately advise their patients and prescribe exercise.

Walking exercise may occur over-ground or on a treadmill. When an individual with a lower-limb amputation is walking over-ground, their right-to-left side walking pattern will be more asymmetrical (uneven) when compared to when they are walking on a treadmill. When walking is more symmetrical side-to-side (even), the patient may have to expend more energy. Energy expenditure can be assessed as the amount of oxygen consumed, which can be obtained while wearing a mask that evaluates the participant's breathing while walking. Among adults with a lower-limb amputation, energy expenditure studies have generally used treadmills to look at energy expenditure. Over-ground versus treadmill conditions, however, are different, and as such, what equals 3 METs (speed, cadence) in each walking condition may vary.

Further, no studies have compared the energy cost of walking in adults who are inactive with a lower-limb amputation to age-, sex-, and body mass index (computed from height and weight) -matched adults without an amputation. While studies have evaluated the impact of aging and limb length of the amputated limb on energy expenditure, few have evaluated modifiable factors that may impact energy expenditure among adults with lower-limb amputation. Similarly, little research has explored modifiable factors that may impact physical activity levels.

The project's goal is to provide knowledge that will improve physical activity prescription for inactive adults with a single, below-the-knee amputation (i.e. transtibial amputation).

Successful completion of the project may provide healthcare providers with (1) a physical activity self-report measure that can be used in clinical practice for patients with a lower-limb amputation, (2) gait speed (mph) for prescribing moderate-intensity over-ground and treadmill walking during the rehabilitation of patients with lower-limb amputations, and (3) cadence (steps/minute), for evaluating and monitoring moderate-intensity physical activity via step activity monitors, for inactive adults with a lower-limb amputation.

Investigators will provide the first objective data that looks at the additional energy expenditure necessary for inactive adults with a lower-limb amputation who are using a prosthesis to walk short-distances as compared to able-bodied adults; this data may be used for the development of future prosthetic components that reduce energy expenditure. Investigators will explore factors that may be linked to energy expenditure and physical activity among adults with and without a lower-limb amputation.

ELIGIBILITY:
Inclusion Criteria (all participants):

* Ages 18-60 years
* Able to read and speak English
* Saltin-Grimby Physical Activity Level of I or II

Inclusion Criteria (individuals with unilateral, transtibial amputations):

* Unilateral, transtibial (below-the-knee) amputation
* Currently wearing a prosthesis with use of an assistive device no greater than a cane
* Wearing prosthetic at least 8 hours per day and inside and outside the home: This criteria will help to ensure that adults are beyond the initial weaning into a prosthetic period and are prosthetic users rather than nonusers.

Inclusion Criteria (controls):

* Pain-free in the legs and low back regions
* Able to walk without an assistive device

Exclusion Criteria:

* Current infections or illnesses that would affect safe participation in the study
* Past medical history of significant cardiovascular disease (e.g. congestive heart failure or previous heart attacks), significant neurological disease (e.g. Parkinson's, Multiple Sclerosis) significant neurological event (e.g. stroke), or major lung condition (e.g. Chronic obstructive pulmonary disease, emphysema)
* Uncontrolled high blood pressure
* Uncontrolled Diabetes Mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Investigators will recruit 22 (males and females) with a unilateral (i.e. single limb), transtibial (i.e. below-the-knee) amputation. Given the prevalence of amputations is greater in males, it is expected that the sample will be predominantly male, but there will not be any inclusion/exclusion criteria related to sex. 20 controls will be recruited as age-, sex-, and body mass index-matched controls for those with a unilateral transtibial amputation who complete the entire study evaluation protocol.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change in gait speed pre- and post-walking tests | immediately before/after
  self-selected and fast speeds obtained with GaitRite

SECONDARY OUTCOMES:
Change in gait symmetry | immediately before/after
  Temporal and spatial gait characteristics obtained with GaitRite

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn M Sions, PhD, PT, DPT, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware STAR Campus, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swaminathan A, Vemulapalli S, Patel MR, Jones WS. Lower extremity amputation in peripheral artery disease: improving patient outcomes. Vasc Health Risk Manag. 2014 Jul 16;10:417-24. doi: 10.2147/VHRM.S50588. eCollection 2014. PMID 25075192
- [Background] Schuch F, Vancampfort D, Firth J, Rosenbaum S, Ward P, Reichert T, Bagatini NC, Bgeginski R, Stubbs B. Physical activity and sedentary behavior in people with major depressive disorder: A systematic review and meta-analysis. J Affect Disord. 2017 Mar 1;210:139-150. doi: 10.1016/j.jad.2016.10.050. Epub 2016 Nov 29. PMID 28033521
- [Background] Shuval K, Leonard T, Drope J, Katz DL, Patel AV, Maitin-Shepard M, Amir O, Grinstein A. Physical activity counseling in primary care: Insights from public health and behavioral economics. CA Cancer J Clin. 2017 May 6;67(3):233-244. doi: 10.3322/caac.21394. Epub 2017 Feb 15. PMID 28198998
- [Background] Tudor-Locke C, Bassett DR Jr. How many steps/day are enough? Preliminary pedometer indices for public health. Sports Med. 2004;34(1):1-8. doi: 10.2165/00007256-200434010-00001. PMID 14715035
- [Background] Klute GK, Berge JS, Orendurff MS, Williams RM, Czerniecki JM. Prosthetic intervention effects on activity of lower-extremity amputees. Arch Phys Med Rehabil. 2006 May;87(5):717-22. doi: 10.1016/j.apmr.2006.02.007. PMID 16635636
- [Background] Halsne EG, Waddingham MG, Hafner BJ. Long-term activity in and among persons with transfemoral amputation. J Rehabil Res Dev. 2013;50(4):515-30. doi: 10.1682/jrrd.2012.04.0066. PMID 23934872
- [Background] Desveaux L, Goldstein RS, Mathur S, Hassan A, Devlin M, Pauley T, Brooks D. Physical Activity in Adults with Diabetes Following Prosthetic Rehabilitation. Can J Diabetes. 2016 Aug;40(4):336-41. doi: 10.1016/j.jcjd.2016.02.003. Epub 2016 Apr 1. PMID 27052673
- [Background] Thyregod M, Bodtger U. Coherence between self-reported and objectively measured physical activity in patients with chronic obstructive lung disease: a systematic review. Int J Chron Obstruct Pulmon Dis. 2016 Nov 25;11:2931-2938. doi: 10.2147/COPD.S116422. eCollection 2016. PMID 27932873
- [Background] Prince SA, Adamo KB, Hamel ME, Hardt J, Connor Gorber S, Tremblay M. A comparison of direct versus self-report measures for assessing physical activity in adults: a systematic review. Int J Behav Nutr Phys Act. 2008 Nov 6;5:56. doi: 10.1186/1479-5868-5-56. PMID 18990237
- [Background] Rowe DA, McMinn D, Peacock L, Buis AW, Sutherland R, Henderson E, Hewitt A. Cadence, energy expenditure, and gait symmetry during music-prompted and self-regulated walking in adults with unilateral transtibial amputation. J Phys Act Health. 2014 Feb;11(2):320-9. doi: 10.1123/jpah.2012-0056. Epub 2013 Jan 30. PMID 23364470
- [Background] Tudor-Locke C, Sisson SB, Collova T, Lee SM, Swan PD. Pedometer-determined step count guidelines for classifying walking intensity in a young ostensibly healthy population. Can J Appl Physiol. 2005 Dec;30(6):666-76. doi: 10.1139/h05-147. PMID 16485518
- [Background] Tudor-Locke C, Rowe DA. Using cadence to study free-living ambulatory behaviour. Sports Med. 2012 May 1;42(5):381-98. doi: 10.2165/11599170-000000000-00000. PMID 22462794
- [Background] Waters RL, Perry J, Antonelli D, Hislop H. Energy cost of walking of amputees: the influence of level of amputation. J Bone Joint Surg Am. 1976 Jan;58(1):42-6. PMID 1249111
- [Background] Tekin L, Safaz Y, Goktepe AS, Yazycyodlu K. Comparison of quality of life and functionality in patients with traumatic unilateral below knee amputation and salvage surgery. Prosthet Orthot Int. 2009 Mar;33(1):17-24. doi: 10.1080/03093640802482542. PMID 19235062
- [Background] Akarsu S, Tekin L, Safaz I, Goktepe AS, Yazicioglu K. Quality of life and functionality after lower limb amputations: comparison between uni- vs. bilateral amputee patients. Prosthet Orthot Int. 2013 Feb;37(1):9-13. doi: 10.1177/0309364612438795. Epub 2012 Jul 24. PMID 22833517
- [Background] Alton F, Baldey L, Caplan S, Morrissey MC. A kinematic comparison of overground and treadmill walking. Clin Biomech (Bristol). 1998 Sep;13(6):434-440. doi: 10.1016/s0268-0033(98)00012-6. PMID 11415818
- [Background] Mattes SJ, Martin PE, Royer TD. Walking symmetry and energy cost in persons with unilateral transtibial amputations: matching prosthetic and intact limb inertial properties. Arch Phys Med Rehabil. 2000 May;81(5):561-8. doi: 10.1016/s0003-9993(00)90035-2. PMID 10807092
- [Background] Lin-Chan SJ, Bilodeau M, Yack HJ, Nielsen DH. The force-driven harmonic oscillator model for energy-efficient locomotion in individuals with transtibial amputation. Hum Mov Sci. 2004 Apr;22(6):611-30. doi: 10.1016/j.humov.2003.12.001. PMID 15063044
- [Background] Esposito ER, Rodriguez KM, Rabago CA, Wilken JM. Does unilateral transtibial amputation lead to greater metabolic demand during walking? J Rehabil Res Dev. 2014;51(8):1287-96. doi: 10.1682/JRRD.2014.06.0141. PMID 25671680
- [Background] Schnall BL, Wolf EJ, Bell JC, Gambel J, Bensel CK. Metabolic analysis of male servicemembers with transtibial amputations carrying military loads. J Rehabil Res Dev. 2012;49(4):535-44. doi: 10.1682/jrrd.2011.04.0075. PMID 22773257
- [Background] Button C, Moyle S, Davids K. Comparison of below-knee amputee gait performed overground and on a motorized treadmill. Adapt Phys Activ Q. 2010 Apr;27(2):96-112. doi: 10.1123/apaq.27.2.96. PMID 20440022
- [Background] Traballesi M, Porcacchia P, Averna T, Brunelli S. Energy cost of walking measurements in subjects with lower limb amputations: a comparison study between floor and treadmill test. Gait Posture. 2008 Jan;27(1):70-5. doi: 10.1016/j.gaitpost.2007.01.006. Epub 2007 Mar 13. PMID 17360186
- [Background] Delbaere K, Hauer K, Lord SR. Evaluation of the incidental and planned activity questionnaire (IPEQ) for older people. Br J Sports Med. 2010 Nov;44(14):1029-34. doi: 10.1136/bjsm.2009.060350. Epub 2009 May 26. PMID 19474003
- [Background] Doma K, Speyer R, Leicht AS, Cordier R. Comparison of psychometric properties between usual-week and past-week self-reported physical activity questionnaires: a systematic review. Int J Behav Nutr Phys Act. 2017 Jan 31;14(1):10. doi: 10.1186/s12966-017-0470-6. PMID 28137268
- [Background] Abel M, Hannon J, Mullineaux D, Beighle A. Determination of step rate thresholds corresponding to physical activity intensity classifications in adults. J Phys Act Health. 2011 Jan;8(1):45-51. doi: 10.1123/jpah.8.1.45. PMID 21297184
- [Background] Harrington DM, Dowd KP, Tudor-Locke C, Donnelly AE. A steps/minute value for moderate intensity physical activity in adolescent females. Pediatr Exerc Sci. 2012 Aug;24(3):399-408. doi: 10.1123/pes.24.3.399. PMID 22971556
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Houghton AD, Taylor PR, Thurlow S, Rootes E, McColl I. Success rates for rehabilitation of vascular amputees: implications for preoperative assessment and amputation level. Br J Surg. 1992 Aug;79(8):753-5. doi: 10.1002/bjs.1800790811. PMID 1393461
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Hafner BJ, Morgan SJ, Askew RL, Salem R. Psychometric evaluation of self-report outcome measures for prosthetic applications. J Rehabil Res Dev. 2016;53(6):797-812. doi: 10.1682/JRRD.2015.12.0228. PMID 28273329
- [Background] Amtmann D, Morgan SJ, Kim J, Hafner BJ. Health-related profiles of people with lower limb loss. Arch Phys Med Rehabil. 2015 Aug;96(8):1474-83. doi: 10.1016/j.apmr.2015.03.024. Epub 2015 Apr 25. PMID 25917819
- [Background] Miller WC, Deathe AB, Speechley M. Psychometric properties of the Activities-specific Balance Confidence Scale among individuals with a lower-limb amputation. Arch Phys Med Rehabil. 2003 May;84(5):656-61. doi: 10.1016/s0003-9993(02)04807-4. PMID 12736877
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Heinemann AW, Magasi S, Bode RK, Hammel J, Whiteneck GG, Bogner J, Corrigan JD. Measuring enfranchisement: importance of and control over participation by people with disabilities. Arch Phys Med Rehabil. 2013 Nov;94(11):2157-65. doi: 10.1016/j.apmr.2013.05.017. Epub 2013 Jun 13. PMID 23769764
- [Background] Heinemann AW, Lai JS, Magasi S, Hammel J, Corrigan JD, Bogner JA, Whiteneck GG. Measuring participation enfranchisement. Arch Phys Med Rehabil. 2011 Apr;92(4):564-71. doi: 10.1016/j.apmr.2010.07.220. Epub 2011 Mar 2. PMID 21367395
- [Background] Linn BS, Linn MW, Gurel L. Cumulative illness rating scale. J Am Geriatr Soc. 1968 May;16(5):622-6. doi: 10.1111/j.1532-5415.1968.tb02103.x. No abstract available. PMID 5646906
- [Background] Gailey RS, Roach KE, Applegate EB, Cho B, Cunniffe B, Licht S, Maguire M, Nash MS. The amputee mobility predictor: an instrument to assess determinants of the lower-limb amputee's ability to ambulate. Arch Phys Med Rehabil. 2002 May;83(5):613-27. doi: 10.1053/apmr.2002.32309. PMID 11994800
- [Background] Buatois S, Miljkovic D, Manckoundia P, Gueguen R, Miget P, Vancon G, Perrin P, Benetos A. Five times sit to stand test is a predictor of recurrent falls in healthy community-living subjects aged 65 and older. J Am Geriatr Soc. 2008 Aug;56(8):1575-7. doi: 10.1111/j.1532-5415.2008.01777.x. No abstract available. PMID 18808608
- [Background] Whitney SL, Wrisley DM, Marchetti GF, Gee MA, Redfern MS, Furman JM. Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther. 2005 Oct;85(10):1034-45. PMID 16180952
- [Background] Horn LB, Rice T, Stoskus JL, Lambert KH, Dannenbaum E, Scherer MR. Measurement Characteristics and Clinical Utility of the Clinical Test of Sensory Interaction on Balance (CTSIB) and Modified CTSIB in Individuals With Vestibular Dysfunction. Arch Phys Med Rehabil. 2015 Sep;96(9):1747-8. doi: 10.1016/j.apmr.2015.04.003. No abstract available. PMID 26550644
- [Background] Gremeaux V, Damak S, Troisgros O, Feki A, Laroche D, Perennou D, Benaim C, Casillas JM. Selecting a test for the clinical assessment of balance and walking capacity at the definitive fitting state after unilateral amputation: a comparative study. Prosthet Orthot Int. 2012 Dec;36(4):415-22. doi: 10.1177/0309364612437904. Epub 2012 Mar 2. PMID 22389424
- [Background] Dite W, Connor HJ, Curtis HC. Clinical identification of multiple fall risk early after unilateral transtibial amputation. Arch Phys Med Rehabil. 2007 Jan;88(1):109-14. doi: 10.1016/j.apmr.2006.10.015. PMID 17207685
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Hess RJ, Brach JS, Piva SR, VanSwearingen JM. Walking skill can be assessed in older adults: validity of the Figure-of-8 Walk Test. Phys Ther. 2010 Jan;90(1):89-99. doi: 10.2522/ptj.20080121. Epub 2009 Dec 3. PMID 19959654
- [Background] Deathe AB, Miller WC. The L test of functional mobility: measurement properties of a modified version of the timed "up & go" test designed for people with lower-limb amputations. Phys Ther. 2005 Jul;85(7):626-35. PMID 15982169
- [Background] Rodjer L, Jonsdottir IH, Rosengren A, Bjorck L, Grimby G, Thelle DS, Lappas G, Borjesson M. Self-reported leisure time physical activity: a useful assessment tool in everyday health care. BMC Public Health. 2012 Aug 24;12:693. doi: 10.1186/1471-2458-12-693. PMID 22920914
- [Background] Devlin M, Pauley T, Head K, Garfinkel S. Houghton Scale of prosthetic use in people with lower-extremity amputations: Reliability, validity, and responsiveness to change. Arch Phys Med Rehabil. 2004 Aug;85(8):1339-44. doi: 10.1016/j.apmr.2003.09.025. PMID 15295762
- [Background] Gailey RS, Wenger MA, Raya M, Kirk N, Erbs K, Spyropoulos P, Nash MS. Energy expenditure of trans-tibial amputees during ambulation at self-selected pace. Prosthet Orthot Int. 1994 Aug;18(2):84-91. doi: 10.3109/03093649409164389. PMID 7991365
- [Background] de Groot V, Beckerman H, Lankhorst GJ, Bouter LM. How to measure comorbidity. a critical review of available methods. J Clin Epidemiol. 2003 Mar;56(3):221-9. doi: 10.1016/s0895-4356(02)00585-1. PMID 12725876
- [Background] Bell JC, Wolf EJ, Schnall BL, Tis JE, Potter BK. Transfemoral amputations: is there an effect of residual limb length and orientation on energy expenditure? Clin Orthop Relat Res. 2014 Oct;472(10):3055-61. doi: 10.1007/s11999-014-3630-x. PMID 24752912
- [Background] Schrack JA, Simonsick EM, Ferrucci L. The relationship of the energetic cost of slow walking and peak energy expenditure to gait speed in mid-to-late life. Am J Phys Med Rehabil. 2013 Jan;92(1):28-35. doi: 10.1097/PHM.0b013e3182644165. PMID 22854908
- [Background] Schrack JA, Simonsick EM, Ferrucci L. The energetic pathway to mobility loss: an emerging new framework for longitudinal studies on aging. J Am Geriatr Soc. 2010 Oct;58 Suppl 2(Suppl 2):S329-36. doi: 10.1111/j.1532-5415.2010.02913.x. PMID 21029063
- [Background] Seefeldt V, Malina RM, Clark MA. Factors affecting levels of physical activity in adults. Sports Med. 2002;32(3):143-68. doi: 10.2165/00007256-200232030-00001. PMID 11839079
- [Background] Moore-Harrison T, Lightfoot JT. Driven to be inactive? The genetics of physical activity. Prog Mol Biol Transl Sci. 2010;94:271-90. doi: 10.1016/B978-0-12-375003-7.00010-8. PMID 21036329
- [Background] Torburn L, Powers CM, Guiterrez R, Perry J. Energy expenditure during ambulation in dysvascular and traumatic below-knee amputees: a comparison of five prosthetic feet. J Rehabil Res Dev. 1995 May;32(2):111-9. PMID 7562650
- [Background] Czerniecki JM, Morgenroth DC. Metabolic energy expenditure of ambulation in lower extremity amputees: what have we learned and what are the next steps? Disabil Rehabil. 2017 Jan;39(2):143-151. doi: 10.3109/09638288.2015.1095948. Epub 2015 Oct 12. PMID 26458225

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03722797/Prot_SAP_000.pdf